CLINICAL TRIAL: NCT01036399
Title: Study of Lenalidomide (Revlimid) in Patients With Relapsed/Refractory Peripheral T-cell Lymphoma (PTCL) Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The EC withdrawn the approval becuase of possible conflicts of interests between our Institute and Supporter (Celgene)
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Pier Luigi Zinzani, Professor, University of Bologna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RV-PTCL-PI-277; EUDRACT 2007-003911-29
Record Dates: First submitted 2009-07-07; First posted 2009-12-21 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-08

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: PTCL
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Revlimid (Experimental): Oral Revlimid is initiated on day 1 of cycle 1at the dose of 25 mg daily for 21 days with 7 days rest (28 day cycle) for a total of 4 cycles.
  After this induction phase, the CR, PR and SD will continue Revlimid with the same schedule for other 8 months.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Oral Lenalidomide is initiated on day 1 of cycle 1at the dose of 25 mg daily for 21 days with 7 days rest (28 day cycle) for a total of 4 cycles.
  Other Names: Revlimid

SUMMARY:
Revlimid is a potent immunomodulatory analogue without the teratogenic effects, which has direct anti-tumor effects, anti-angiogenic and both anti-inflammatory and T-cell costimulatory properties. Both preclinical and clinical data indicate its efficacy solid tumor and multiple myeloma including advanced/refractory stages with its role in enhancing host antitumor immunity that provided the rationale to use in patients with PTCL.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologic diagnosis of PTCL according to the WHO-REAL classification;
* Age > 18 years;
* Relapsed (³1) or refractory to conventional chemotherapy/radiotherapy;
* Stage I-IV according to the Ann Arbor staging System;
* Performance status <2;
* Adequate bone marrow reserve: platelets >50 x 10(9)/L, absolute neutrophil count
* (ANC) > 1.0 x 10(9)/L, hemoglobin >8 g/d;
* Normal renal and hepatic functions;
* Negative HIV, HCV, and HBV status;
* Informed consent prior to registration on study

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 28 days of baseline.
* Known hypersensitivity to thalidomide.
* The development of erythema if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Any prior use of lenalidomide.
* Concurrent use of other anti-cancer agents or treatments.
* Known positive for HIV or infectious hepatitis, type A, B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-11; Primary Completion 2009-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility of Revlimid as salvage treatment in PTCL | 12 months

SECONDARY OUTCOMES:
To assess the overall response rate (CR and PR) of PTCL receiving REVLIMID; To assess the Tumor Control Rate (TCR); To assess the duration of response; To assess the quality of life. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute Of Hematology "Seràgnoli", Bologna, Italy

REFERENCES:
- [Derived] Zinzani PL, Pellegrini C, Broccoli A, Stefoni V, Gandolfi L, Quirini F, Argnani L, Berti E, Derenzini E, Pileri S, Baccarani M. Lenalidomide monotherapy for relapsed/refractory peripheral T-cell lymphoma not otherwise specified. Leuk Lymphoma. 2011 Aug;52(8):1585-8. doi: 10.3109/10428194.2011.573031. Epub 2011 Apr 19. No abstract available. PMID 21504290